CLINICAL TRIAL: NCT04907812
Title: The Role of Tranexamic Acid in Reducing Post Operative Hand Edema After Hand and Wrist Surgery (THAW): A Prospective, Randomized Controlled, Double-Blinded Pilot Study
Brief Title: The Role of Tranexamic Acid in Reducing Post Operative Hand Edema After Hand and Wrist Surgery
Acronym: THAW
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruby Grewal (Other)
Responsible Party: Sponsor-Investigator, Ruby Grewal, Co-director of the clinical research lab within the Roth | McFarlane Hand and Upper Limb Center (HULC), London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116724
Record Dates: First submitted 2021-04-06; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Hand Injuries and Disorders; Distal Radius Fracture; Dupuytren Contracture
Keywords: swelling; edema; distal radius fracture; dupuytren; Tranexamic Acid
MeSH Terms: conditions — Hand Injuries; Disease; Wrist Fractures; Dupuytren Contracture; Edema | interventions — Tranexamic Acid; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: A Prospective, Randomized Controlled, Double-Blinded Pilot Study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic Acid (TXA) (Experimental): Patients in the TXA arm will receive 1 gram dose of intravenous (IV) tranexamic acid mixed with 50cc 0.9% sodium chloride before their surgery and 1 gram dose of intravenous (IV) tranexamic acid mixed with 50cc 0.9% sodium chloride 3-6 hours after the first dose on the day of their surgery
  Interventions: Drug: Tranexamic acid; Procedure: Surgery
- Standard of Care (SOC) (Placebo Comparator): Patients in the (SOC) arm will receive 50cc of IV Placebo (standard intravenous normal saline fluid - 0.9% sodium chloride) before their surgery and 50cc of IV Placebo (standard intravenous normal saline fluid - 0.9% sodium chloride) 3-6 hours after the first dose on the day of their surgery
  Interventions: Procedure: Surgery

INTERVENTIONS:
Drug: Tranexamic acid — Patients will receive 1 gram dose of intravenous (IV) tranexamic acid mixed with 50cc 0.9% sodium chloride before your surgery and 1 gram dose of intravenous (IV) tranexamic acid mixed with 50cc 0.9% sodium chloride 3-6 hours after your first dose on the day of your surgery
  Arms: Tranexamic Acid (TXA)
Procedure: Surgery — This will include regional anaesthesia, tourniquet inflation to 250mmHg and perioperative antibiotics. At the conclusion of the procedure hemostasis will be achieved followed by standard closure technique. There will be three separate surgical groups that will undergo the outlined study protocol: 1) Distal radius fractures will be treated with open reduction from a volar approach only technique 2) Mild dupuytren's: a. Low: i. MCP joints <50 contracture ii. PIP joints <40 contracture b. 1-2 fingers involved 3) Severe dupuytren's a. High: i. MCP joints >50 degree contracture ii. PIP Joints >40 degrees contracture b. >2 fingers involved

SUMMARY:
Hand edema following hand surgery is a common yet devastating side effect that can lead to early stiffness, prolonged rehabilitation and diminished function. These factors can reduce a patient's quality of life; mounting to an overall delay in recovery, return to work and daily activities. Conventional edema therapy includes cryotherapy, external compression, active and passive exercises and various types of massage. However, there is little evidence to suggest these modalities are effective. Tranexamic acid (TXA) is an antifibrinolytic that has been used in surgical disciplines for decades to aid in reducing intraoperative blood loss and consequent transfusions. Recently, the use of TXA for curbing post-operative edema and ecchymosis has shown promising results, however, its use in hand surgery has not been studied.

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years old undergoing distal radius fracture open reduction and internal fixation through a volar approach at St. Joseph's hospital in London, Ontario
* All patients >18 years old undergoing open fasciectomy for Dupuytren's disease at St. Joseph's hospital in London, Ontario

Exclusion Criteria:

* Revision surgery
* Distal radius fractures treated with additive or alternative approaches and fixation to the volar approach
* Known history of lymphedema or lymph node dissection on either upper extremity
* Known allergic reaction to TXA
* Cardiovascular problems (history of myocardial infraction, angina, and atrial fibrillation)
* Cerebrovascular conditions (history of previous stroke)
* Thromboembolic disorders (history of deep vein thrombosis [DVT] or pulmonary embolism [PE]), clotting disorders)
* Known seizure disorder
* Currently on dialysis
* Current pregnancy or breastfeeding
* Current use of hormone contraception
* Unable to read consent and patient surveys related to the study in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to protocol | 12 weeks
  Assess number of patients who receive hand volume measurements at all designated time intervals. The outcome goal will be 90%
Treatment Completion Rate | 12 weeks
  Asses proportion of patients who correctly receive the intervention as per the protocol. The outcome goal will be 90%
Retention Rate | 12 weeks
  Proportion of participants to complete the study protocol and associated follow up. The outcome goal will be an 80% retention rate
Recruitment rate | 12 weeks
  Number of patients recruited to the study per month. The outcome goal will be 5 patients per month

SECONDARY OUTCOMES:
Hand volume | 12 weeks
  Hand volume will be assessed using two validated methods; water displacement and figure of eight measurement.
Patient-reported pain scores | 12 weeks
  Patient Reported Wrist and Hand Evaluation (PRWHE). The PRWHE allows patients to rate their levels of hand and wrist pain and disability. It is rated on a 0-100 scale. A higher score in the scale denotes a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Lawson Health Research Institute, London, Ontario, Canada